CLINICAL TRIAL: NCT03595306
Title: Human Gut Microbiota and Prebiotic Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00087214
Record Dates: First submitted 2018-07-11; First posted 2018-07-23 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy Gut Microbiota

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prebiotic A (Experimental)
  Interventions: Dietary Supplement: Prebiotic A - inulin; Dietary Supplement: Prebiotic B - galactooligosaccharides(GOS); Dietary Supplement: Prebiotic C - wheat dextrin
- Prebiotic B (Experimental)
  Interventions: Dietary Supplement: Prebiotic A - inulin; Dietary Supplement: Prebiotic B - galactooligosaccharides(GOS); Dietary Supplement: Prebiotic C - wheat dextrin
- Prebiotic C (Experimental)
  Interventions: Dietary Supplement: Prebiotic A - inulin; Dietary Supplement: Prebiotic B - galactooligosaccharides(GOS); Dietary Supplement: Prebiotic C - wheat dextrin

INTERVENTIONS:
Dietary Supplement: Prebiotic A - inulin — Pre-weighed packages will be given twice daily for 5 days.
Dietary Supplement: Prebiotic B - galactooligosaccharides(GOS) — Pre-weighed packages will be given twice daily for 5 days.
Dietary Supplement: Prebiotic C - wheat dextrin — Pre-weighed packages will be given twice daily for 5 days.

SUMMARY:
This study is designed to examine the shift in gut microbiota and their metabolism after consumption of a dietary supplement (prebiotic) by healthy participants. The investigators will provide participants with a panel of over the counter prebiotics and monitor their gut microbiome response in stool. All prebiotics will be commercially available, over-the-counter food, food additives, or dietary supplements, without any known market-use adverse effects beyond minimal discomfort.

ELIGIBILITY:
Inclusion Criteria:

* Provide Stool Samples at no risk to yourself

Exclusion Criteria:

* No oral antibiotic treatments within previous 1 month
* No known allergy to milk products or lactose intolerance
* no known allergy to wheat or gluten intolerance
* no history of irritable bowel syndrome
* no history of inflammatory bowel disease
* no history of type-2 diabetes
* no history of chronic kidney disease or reduced kidney function
* no current intestinal obstructions
* no current untreated colorectal cancer
* not currently pregnant or breastfeeding

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-05-19 (Actual); Study Completion 2019-05-19 (Actual)

PRIMARY OUTCOMES:
change in levels of SCFAs in stool samples | Baseline and 6 weeks

SECONDARY OUTCOMES:
change in levels of cytokines in stool samples | Baseline and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence David, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States